CLINICAL TRIAL: NCT04791553
Title: A Phase 1, Open-Label, Pharmacokinetic, Safety and Tolerability Study of a Single Oral Dose of Cenobamate (YKP3089) in Subjects With Normal Hepatic Function and Subjects With Severe Hepatic Impairment
Brief Title: Safety Study of Cenobamate in Subjects With Normal Hepatic Function and Subjects With Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: YKP3089C038
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — Cenobamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal Hepatic Function (Experimental): Group 1 single oral dose of 200 mg (2 x 100 mg tablet) cenobamate given to Matching healthy subjects with normal hepatic function
  Interventions: Drug: Cenobamate
- Hepatic Impairment (Experimental): Group 2 single oral dose of 200 mg (2 x 100 mg tablet) cenobamate given to subjects with severe hepatic impairment
  Interventions: Drug: Cenobamate

INTERVENTIONS:
Drug: Cenobamate — Cenobamate (YKP3089) is a small molecule approved in the United States (US) for the treatment of partial onset seizures (POS) in adult patients.
  Other Names: YKP3089

SUMMARY:
This study is designed investigate the effect of severe hepatic impairment on the pharmacokinetics (PK) of cenobamate.

DETAILED DESCRIPTION:
This is a Phase 1, multi-center, open-label, non-randomized, parallel group PK and safety study of a single oral dose of cenobamate in male and female subjects with normal hepatic function (Group 1, n = 8) and those with severe hepatic impairment (Group 2, n = 8).

The study consists of a 28-day screening period, followed by single dose administration of cenobamate (200mg) on Day 1, an assessment period of 35 days and follow-up visit. All subjects will be confined to the clinical site from Day -1 (the day before dosing) until Day 5. Outpatient visits will be performed regularly until Day 35. The follow-up visit will occur on Day 40 (±1 day).

ELIGIBILITY:
Inclusion Criteria:

* All Subjects

  1. Able to understand and willing to sign the ICF and able to comply with the study restrictions
  2. Adult male or female subjects age 18 to 75 years, inclusive, at the time of informed consent
  3. BMI 18.0 - 35.0 kg/m2, inclusive, where BMI (kg/m2) = body weight (kg) / height2 (m2) at Screening
  4. Female subjects of childbearing potential willing to use an acceptable form of birth control, as outlined in Section 12.1.9
  5. Male subjects with female partners of childbearing potential may be enrolled if they, use an acceptable form of birth control, as outlined in Section 12.1.9

Hepatically-impaired Subjects (in addition)

1. Diagnosis of cirrhosis due to parenchymal liver disease, which is confirmed and documented by at least one of the following: medical history, physical examination, hepatic ultrasound, computed tomography (CT) scan, magnetic resonance imaging (MRI), and/or liver biopsy
2. Stable hepatic impairment (Child-Pugh score consistent with severe hepatic impairment), defined as no clinically significant change in disease status, as judged by the Investigator

Healthy Subjects (in addition)

1. Subjects with normal hepatic function as judged by the Investigator
2. Judged to be in good health in the opinion of the Investigator on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality (including a physical examination, medical history, ECG, vital signs, and the results of biochemistry, coagulation and hematology tests and urinalysis carried out at Screening) or Subject has a stable disease (e.g., hypertension, hyperlipidemia, diabetes mellitus, hyperthyreosis) under medical control (i.e., adequate treatment), and does not show clinically relevant abnormalities that are not in line with the underlying disease

Exclusion Criteria:

* All subjects

  1. Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at Screening that the Investigator judges as likely to interfere with the objectives of the trial or the safety of the volunteer except for conditions associated with hepatic impairment in subjects with compromised hepatic function (Group 2)
  2. Any surgical or medical condition that may significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study
  3. History of or present epileptic episodes or suicidal attempts
  4. Documented congenital QT syndrome
  5. Corrected QT interval (QTc) using Fridericia correction (QTcF) at Screening or predose > 450 ms or < 350 ms
  6. Unstable ischemic heart disease or severe heart failure (New York Heart Association Class III or IV)
  7. Uncontrolled treated/untreated hypertension (defined as a mean of 3 repeated measurements for systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 105 mmHg); current or documented history of repeated clinically significant hypotension
  8. Primary biliary cirrhosis
  9. Subject has a history of any serious drug-induced hypersensitivity reaction (including, but not limited to, Stevens Johnson syndrome, toxic epidermal necrolysis, or Drug Reaction with Eosinophilia and Systemic Symptoms [DRESS]) or any drug-related rash requiring hospitalization
  10. History of AED-associated rash that involved conjunctiva or mucosae
  11. History of more than one non-serious drug-related hypersensitivity reaction that required discontinuation of the medication
  12. Known hypersensitivity or previous intolerance to cenobamate or any of its excipients
  13. History of cancer (judged not to be in full remission) or presence of cancer (except basal cell skin cancer or squamous cell skin cancer) as judged by the Investigator
  14. Acute illness within 14 days prior to study drug administration unless mild in severity and approved by the Investigator and Sponsor's medical representative
  15. Active infection of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)
  16. Presence of active infection requiring antibiotics
  17. Concomitant use of medications known to be linked with DRESS syndrome (including carbamazepine, lamotrigine, phenytoin, any sulfonamide [e.g., sulfasalazine, dapsone, sulfamethoxazole], minocycline and nevirapine, abacavir) should be excluded at least 4 weeks prior to dosing and up to 4 weeks post cenobamate dosing
  18. Use of any prescription or non-prescription drugs, including over-the-counter medication, non-routine vitamins and herbal products within 2 weeks prior to study drug administration unless discussed and agreed with the Sponsor's medical representative in writing (Medication used to treat TEAEs does not lead to a compulsory exclusion of subjects)
  19. Ingestion of alcohol within 72 hours prior to study drug administration and during inhouse period. Outside the in-house period, regular alcohol consumption below 24 units for males and 17 units for females per week (1 unit equals 250 mL of beer, 75 mL of wine or 25 mL of spirits) is allowed
  20. Active smokers within the last 6 months
  21. Consumption of an average of more than 5 servings (240 mL per serving) per day of coffee, cola, or other caffeinated beverage before screening. Subjects may not consume any caffeinated beverages from 48 hours prior to dosing until the end of the in-house stay on Day 5.
  22. Participation in a clinical study involving administration of either an investigational or a marketed drug within 2 months or 7 half-lives (whichever is longer) before Screening
  23. Donation or loss of more than 450 mL blood during the 3 months before the start of Screening
  24. Female subjects who are pregnant, nursing, or planning to become pregnant during the study
  25. Clinically significant renal disease (creatinine clearance [CLCr] < 60 mL/min as calculated by the Cockcroft-Gault formula at Screening)
  26. Positive serology for human immunodeficiency virus antibodies (anti-HIV-1/2) at Screening.
  27. Positive urine drug screen (if not due to concomitant medication) or alcohol breath test at Screening and/or Day -1
  28. Legal incapacity or limited legal capacity
  29. Consumption of grapefruit or grapefruit-containing products within 48 hours before Study Day 1 and during the PK sampling period.

Hepatically-impaired Subjects (in addition)

1. History of esophageal bleeding within the last 3 months prior to study drug administration.
2. Severe hepatic encephalopathy (Grade > 2) or degree of central nervous system (CNS) impairment which the Investigator considers sufficiently serious to interfere with the informed consent, the conduct, the completion, or the results of this trial, or constitutes an unacceptable risk to the subject
3. Has had clinical exacerbation of liver disease within 14 days before study drug administration (e.g., abdominal pain, ascites, nausea, vomiting, anorexia, fever, or worsening of laboratory results related to hepatic function)
4. Has evidence of acute viral hepatitis within 1 month before Day -1
5. Has evidence of severe or acute renal failure
6. History of drug or alcohol abuse within 3 months prior to dosing
7. Any significant change in chronic treatment medication within 14 days before inclusion
8. Any medical condition other than hepatic impairment which might alter the drug metabolism
9. Have used any drugs known to significantly affect hepatic metabolism within 28 days, or is unable or unwilling to forgo the use of such products throughout the study
10. Has evidence of hepato-renal syndrome
11. Have acute, fulminant alcoholic hepatitis, determined either clinically or by histology, hepatoma or metastatic disease of the liver
12. History of liver transplantation
13. Advanced ascites and ascites which require emptying and albumin supplementation, as judged by the Investigator
14. Hemoglobin concentration < 105 g/L

Healthy Subjects (in addition)

1. Any clinically unstable, uncontrolled medical condition, which in the opinion of the Investigator would preclude the subject participation to the study
2. Positive serology for HBsAg or anti-HCV
3. History of any illness or condition that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject
4. Illness within 5 days before the start of study drug dosing ("illness" is defined as an acute [serious or non-serious] condition [e.g., the flu or the common cold])
5. History of drug abuse within the last 2 years prior to study drug administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Cmax | 40 days
  Maximum observed plasma concentration of cenobamate
Area Under the Concentration Curve to last measurable concentration | 40 days
  AUC from the time of dosing to the time of the last measurable concentration of cenobamate
Area Under the Concentration Curve from 0 to infinity | 40 days
  AUC from time 0 extrapolated to infinity

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 40 days
  To evaluate the safety and tolerability of cenobamate (Oral Dose of 2x100 mg tablets) administered to matching groups with normal and impaired hepatic function incidence of treatment-emergent adverse events will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Laramy, PhD, PharmD, Study Chair — SK Life Science, Inc.
Locations (2):
- Centrum Badan Klinicznych Piotr Napora lekarze sp.p.,, Wroclaw, Poland
- Summit Clinical Research s.r.o., Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No